CLINICAL TRIAL: NCT00984737
Title: Newly Diagnosed Hyperglycemia and Stress Hyperglycemia in a Coronary Intensive Care Unit
Brief Title: Hyperglycemia in a Coronary Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Purpose: Diagnostic
Other Study IDs: KA07/101
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus; Hyperglycemia; Blood Glucose; Myocardial Ischemia
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Myocardial Ischemia | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Insulin — Capillary glucose measurements of Group 2 and Group 3 will be performed during hospitalization and will be treated when they are over 180mg/dl.
  Short acting oral anti-diabetic drugs will be given to patients who refuse insulin injection.

SUMMARY:
Newly diagnosed hyperglycemia (NDH) and stress hyperglycemia (SH) during acute illness is reported as a non-physiological condition in hospitals. The investigators aim is to determine the rate of NDH and SH among cases admitted to coronary ICU with acute coronary disease and to inquire the relationship of SH with disease severity and functional outcomes such as longevity of ICU stay.

DETAILED DESCRIPTION:
Patients with acute coronary heart disease admitted to the emergency room will be recruited consecutively. Admission plasma glucose (APG) and fasting plasma glucose (FPG); the first morning after admission, measurements will be obtained and each participant will be subjected to capillary glucose measurement (CGM) every six hours within the first day.

Patients will be separated into 4 groups:

GROUP 1: Normoglycemic cases GROUP 2: Newly diagnosed hyperglycemic cases Group 2a: Unrecognized diabetes, hbA1c: >6.0% Group 2b: Stress hyperglycemia <6.0%. GROUP 3: Known diabetes Age, gender, co-morbidities on admission, adverse outcomes in hospital, duration of stay in coronary ICU, deaths, drugs, and glucose levels will be all recorded.

Throughout the hospital stay of Group 2 and Group 3, CGMs were performed and treated when necessary (target glucose<180mg/dl).

Acute Physiology and Chronic Health Evaluation II (APACHE-II); a severity of disease classification system was used for each case.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute coronary syndrome (non ST segment elevation)and myocardial infarction admitted to coronary ICU only via emergency room

Exclusion Criteria:

* Patients admitted to coronary ICU from other hospital wards
* Patients with any disease that will need drugs that may interfere with blood glucose negatively (mannitol, glucocorticoids, vasopressor agents, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence of newly diagnosed hyperglycemia in coronary ICU.

SECONDARY OUTCOMES:
To search for the cases with stress hyperglycemia and inquire its relationship with disease severity and functional outcomes, such as longevity of ICU stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Faculty of Medicine, Adana Medical Center, Adana, Turkey (Türkiye)

REFERENCES:
- [Result] Umpierrez GE, Isaacs SD, Bazargan N, You X, Thaler LM, Kitabchi AE. Hyperglycemia: an independent marker of in-hospital mortality in patients with undiagnosed diabetes. J Clin Endocrinol Metab. 2002 Mar;87(3):978-82. doi: 10.1210/jcem.87.3.8341. PMID 11889147
- [Result] Norhammar AM, Ryden L, Malmberg K. Admission plasma glucose. Independent risk factor for long-term prognosis after myocardial infarction even in nondiabetic patients. Diabetes Care. 1999 Nov;22(11):1827-31. doi: 10.2337/diacare.22.11.1827. PMID 10546015
- [Result] McCowen KC, Malhotra A, Bistrian BR. Stress-induced hyperglycemia. Crit Care Clin. 2001 Jan;17(1):107-24. doi: 10.1016/s0749-0704(05)70154-8. PMID 11219223
- [Result] Capes SE, Hunt D, Malmberg K, Gerstein HC. Stress hyperglycaemia and increased risk of death after myocardial infarction in patients with and without diabetes: a systematic overview. Lancet. 2000 Mar 4;355(9206):773-8. doi: 10.1016/S0140-6736(99)08415-9. PMID 10711923
- [Derived] Ertorer ME, Haydardedeoglu FE, Erol T, Anaforoglu I, Binici S, Tutuncu NB, Sezgin A, Demirag NG. Newly diagnosed hyperglycemia and stress hyperglycemia in a coronary intensive care unit. Diabetes Res Clin Pract. 2010 Oct;90(1):8-14. doi: 10.1016/j.diabres.2010.05.023. Epub 2010 Jul 31. PMID 20674059